CLINICAL TRIAL: NCT02616471
Title: Effect of High Cheese Consumption on Metabolic Syndrome Risk Factors in a Metabolically Vulnerable Population
Brief Title: Effect of High Cheese Consumption on Metabolic Syndrome Risk Factors
Acronym: Osterix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other); Dairy Research Institute (Other); Dairy Farmers of Canada (Other); Centre National Interprofessionel de l'Economie Laitière (Other); Dairy Australia (Industry); Nederlandse Zuivel Organisatie (Other)
Responsible Party: Principal Investigator, Arne Astrup, Prof., MD, Head of Department, Department of Nutrition, Exercise and Sports, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B306
Record Dates: First submitted 2014-01-20; First posted 2015-11-30 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Metabolic Syndrome
Keywords: Cheese; Dairy; Saturated fat; Blood lipid concentrations; Lipoprotein particle size; Metabolic Syndrome; Insulin sensitivity; Blood glucose concentrations
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-fat cheese (HFC) group (Experimental): The subjects in the HFC group will be supplied with equal amounts of two types of regular/high fat cheeses. The cheeses are normal-fat Danbo (Riberhus, 25% fat, Arla, DK) and normal-fat Cheddar (Sharp Cheddar, 32% fat, Cabot, US).
  No further dairy and cheese consumption is allowed
  Interventions: Dietary Supplement: High-fat cheese
- Low-fat cheese (LFC) group (Experimental): The subjects in the LFC group will be supplied with equal amounts of two types of reduced/low fat cheeses. The cheeses are reduced-fat Danbo(Cheasy, 13% fat, Arla, DK) and reduced-fat Cheddar (Sharp Light Cheddar, 16% fat, Cabot, US). No further dairy/cheese consumption is allowed.
  Interventions: Dietary Supplement: Low-fat cheese
- No-cheese/carbohydrate group (CTR) (Active Comparator): For subjects in the CTR group, cheese is replaced by simple and starchy carbohydrates in jam and white bread, which will be supplied by the department. The daily energy and sodium contents will be matched to those of the cheese in the HFC group. No dairy/cheese consumption is allowed.
  Interventions: Dietary Supplement: No-cheese/carbohydrate

INTERVENTIONS:
Dietary Supplement: High-fat cheese
  Arms: High-fat cheese (HFC) group
Dietary Supplement: Low-fat cheese
  Arms: Low-fat cheese (LFC) group
Dietary Supplement: No-cheese/carbohydrate
  Arms: No-cheese/carbohydrate group (CTR)

SUMMARY:
The overall aim of the present research project is to examine whether consumption of high daily amounts of cheese, both high-fat and low-fat, affects risk markers of disease in a study population of men and women with metabolic syndrome risk factors.

It will be explored whether high-fat and/or low-fat cheese consumption can be regarded healthy to consume for at-risk populations (assessed by within-group comparisons from baseline values) and if low-fat or non-fat alternatives to high-fat cheese should continue to be recommended (assessed by between-group comparisons).

In addition, it will be assessed if cheese consumption affects women and men differently as suggested by observational data. The present research project will examine the health effects of cheese as a food product per se and not as a sum of single nutrients, knowing that the single components of cheese cannot be adequately placebo-matched. A relatively high daily intake of high-fat cheese will be compared to a similar intake of low-fat cheese and with a carbohydrate control.

ELIGIBILITY:
Inclusion Criteria:

Men or women

Age 18-70

Waist circumference > 80 cm for women / > 94 cm for men

Plus at least one additional established risk factor for the metabolic syndrome using the following criteria:

* Elevated BP (Systolic BP > 130 mmHg and/or diastolic BP > 85 mmHg);
* Elevated triglycerides (>1.7 mmol/l);
* Reduced HDL-C (<1.0 mmol/l for men and < 1.3 mmol/l for women);
* Elevated fasting glucose (> 5.6 mmol/l). BMI 18.5 - 35 kg/m2

Exclusion Criteria:

Chronic diseases (known diabetes; cardiovascular disease; other chronic diseases which could affect the results of the present study)

Milk allergy

Use of dietary supplements incl. multivitamins (2 months before and during the entire study period)

>10 hours of strenuous physical activity per week

Use of prescription medicine which could affect the results of the present study including systemic glucocorticoids or medicine which have interactions with the intervention products (safety)

Drug or alcohol abuse

Blood donation <1 month before study commencement and during study period

Simultaneous participation in other clinical studies

Pregnant or lactating women, or women who are planning to become pregnant within the next 6 months.

Inability to comply with the procedures required by the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in LDL cholesterol from baseline to post-intervention | week 1 and week 12
  fasting, mmol/l

SECONDARY OUTCOMES:
Blood lipid concentrations | week 1 and week 12
  Total and HDL cholesterol - fasting (mmol/l) Triglycerides - fasting (mmol/l)
Particle size | week 1 and week 12
  HDL, VLDL and LDL particle size (by NMR)
Anthropometry | 5 times during the 12-week intervention
  Hip circumference (cm) Waist circumference (cm) Weight (kg)
Blood pressure (BP) | 3 time during the 12-week intervention
  Systolic BP (mmHG) Diastolic BP (mmHG)
Insulin sensitivity | week 1 and week 12
  Plasma glucose - fasting (mmol/l) Plasma insulin - fasting (mmol/l)
Inflammation | week 1 and week 12
  Serum C-reactive protein - fasting (mmol/l)
Postprandial markers of lipid metabolism | week 12
  Measurements in a sub-group
Postprandial markers of glucose metabolism | week 12
  Measurements in a sub-group
Postprandial appetite sensation (by VAS) | week 12
  Measurements in a sub-group

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof, MD, Principal Investigator — Head of Department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sport, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Raziani F, Tholstrup T, Kristensen MD, Svanegaard ML, Ritz C, Astrup A, Raben A. High intake of regular-fat cheese compared with reduced-fat cheese does not affect LDL cholesterol or risk markers of the metabolic syndrome: a randomized controlled trial. Am J Clin Nutr. 2016 Oct;104(4):973-981. doi: 10.3945/ajcn.116.134932. Epub 2016 Aug 24. PMID 27557654